CLINICAL TRIAL: NCT04394611
Title: Analysis of Some Heavy Metals and Some Vitamins Levels in Maternal Samples, Fetal Samples and Breast Milk for Fetal Growth Restriction.
Brief Title: Metals and in Fetal Growth Restriction
Acronym: FGR&metals
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cengiz Gokcek Women's and Children's Hospital (Other)
Responsible Party: Principal Investigator, Ali Ovayolu, Principal Investigator, Cengiz Gokcek Women's and Children's Hospital
Other Study IDs: CengizGWCH6
Record Dates: First submitted 2020-05-10; First posted 2020-05-19 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Fetal Growth Restriction
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — maternal plasma/urine/hair, cord plasma, placenta and breast milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fetal Growth Restriction (FGR): FGR will be defined as an estimated fetal weight (grams) less than the 10th percentile for gestational age. Hadlock I formula will be used to calculating estimated fetal weight percentiles
  Interventions: Other: Obstetric ultrasound- doppler examination
- Control: healthy pregnancies will be selected for the control group.
  Interventions: Other: Obstetric ultrasound- doppler examination

INTERVENTIONS:
Other: Obstetric ultrasound- doppler examination — Obstetric ultrasound- doppler examination and fetal- maternal assessment Tin (Sn), manganese (Mn), Vanadium (V), Magnesium (Mg), cobalt (Co), nickel (Ni), arsenic (As), chromium (Cr), cadmium (Cd), lead (Pb), mercury (Hg), antimony (Sb), aluminum (Al), zinc (Zn), copper (Cu), selenyum (Se), iron (Fe), vitamin D, vitamin A, vitamin B12 and folate concentrations measurements
  Other Names: metals measurements

SUMMARY:
Introduction: Intrauterine fetal growth restriction (FGR) is a condition in which the fetus does not realize its growth potential in the uterus. Heavy metals important pollutants produced from anthropogenic activities, has been suggested to be embryotoxic and fetotoxic in a lot of studies. However, the causes of fetal growth restriction are little known and heavy metals merit further investigation. The investigators will be tested whether fetal growth restriction was associated with exposure to these metals/vitamins.

Methods: This study was designed to determine maternal plasma/urine/hair, cord plasma, placenta and breast milk tin (Sn), manganese (Mn), Vanadium (V), Magnesium (Mg), cobalt (Co), nickel (Ni), arsenic (As), chromium (Cr), cadmium (Cd), lead (Pb), mercury (Hg), antimony (Sb), aluminium (Al), zinc (Zn), copper (Cu), selenium (Se), iron (Fe), vitamin D, vitamin A, vitamin B12 and folate concentrations in women with FGR (n=55) compared to those of volunteer healthy pregnant women (n=55). These heavy metals concentrations measured using inductively coupled plasma-mass spectrometry were compared.

DETAILED DESCRIPTION:
This observational case-control study will be conducted at the Department of Obstetrics and Gynecology, Cengiz Gokcek Public Hospital, Gaziantep, Turkey, between May 2020 and February 2021. The protocol was approved by the Ethics Committee for Clinical Research of Gaziantep University (reference no: 2020/131). The study strictly will be adhered to the principles of the Declaration of Helsinki. All subjects will be included in the study gave oral and written informed consent. FGR was defined as an estimated fetal weight (grams) less than the 10th percentile for gestational age. Hadlock I formula were used to calculating estimated fetal weight percentiles. Every woman in the study population will be undergone obstetric ultrasound/doppler examination and fetal-maternal assessment will be carried out. Then, this study will be determined maternal plasma/urine/hair, cord plasma, placenta and breast milk tin (Sn), manganese (Mn), Vanadium (V), Magnesium (Mg), cobalt (Co), nickel (Ni), arsenic (As), chromium (Cr), cadmium (Cd), lead (Pb), mercury (Hg), antimony (Sb), aluminium (Al), zinc (Zn), copper (Cu), selenium (Se), iron (Fe), vitamin D, vitamin A, vitamin B12 and folate concentrations in women with FGR (n=55) compared to those of volunteer healthy pregnant women (n=55).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women complicated with fetal growth restriction
* healthy pregnancy
* singleton pregnancy

Exclusion Criteria:

1. pregnant women with any systemic condition (such as chronic hypertension, renal disease and )
2. Women who have dyed their hair in the last 9 months
3. history of using any medication
4. Presence of gestational hypertension or gestational diabetes
5. drug user
6. patients who had fetal congenital abnormalities or genetic syndromes
7. multiple-gestation pregnancies
8. intrauterine fetal death

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnancy
Study Population: The investigators consecutively will be recruited 55 subjects with Fetal growth restriction, and 55 healthy pregnancies will be selected for the control group.
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2020-05-30 (Actual); Primary Completion 2021-11-28 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
measurements of metals (µg/L) and vitamins concentrations for both groups | 10 day
  The primary outcome in these analyses will measure tin (Sn), manganese (Mn), Vanadium (V), Magnesium (Mg), cobalt (Co), nickel (Ni), arsenic (As), chromium (Cr), cadmium (Cd), lead (Pb), mercury (Hg), antimony (Sb), aluminium (Al), zinc (Zn), copper (Cu), selenium (Se), and iron (Fe) concentrations in FGR group and control group. Moreover, the other primary outcome in these analyses will also measure vitamin D, vitamin A, vitamin B12 and folate concentrations in FGR group and control group.

SECONDARY OUTCOMES:
compare the neonatal outcomes for both groups | 1 day
  The secondary outcome in these analyses will compare composite neonatal outcome (APGAR scores, weight, length, head circumference, abdominal circumference, placental weight and NICU admission) in FGR group and control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Cengiz Gokcek Women's and Child's hospital, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Xiong YW, Zhu HL, Nan Y, Cao XL, Shi XT, Yi SJ, Feng YJ, Zhang C, Gao L, Chen YH, Xu DX, Wang H. Maternal cadmium exposure during late pregnancy causes fetal growth restriction via inhibiting placental progesterone synthesis. Ecotoxicol Environ Saf. 2020 Jan 15;187:109879. doi: 10.1016/j.ecoenv.2019.109879. Epub 2019 Oct 31. PMID 31677567
- [Result] Eroglu H, Turgal M, Senat A, Karakoc G, Neselioglu S, Yucel A. Maternal and fetal thiol/disulfide homeostasis in fetal growth restriction. J Matern Fetal Neonatal Med. 2021 May;34(10):1658-1665. doi: 10.1080/14767058.2019.1646239. Epub 2019 Aug 5. PMID 31327276
- [Result] Gordijn SJ, Beune IM, Thilaganathan B, Papageorghiou A, Baschat AA, Baker PN, Silver RM, Wynia K, Ganzevoort W. Consensus definition of fetal growth restriction: a Delphi procedure. Ultrasound Obstet Gynecol. 2016 Sep;48(3):333-9. doi: 10.1002/uog.15884. PMID 26909664
- [Result] Jiang M, Li Y, Zhang B, Zhou A, Zheng T, Qian Z, Du X, Zhou Y, Pan X, Hu J, Wu C, Peng Y, Liu W, Zhang C, Xia W, Xu S. A nested case-control study of prenatal vanadium exposure and low birthweight. Hum Reprod. 2016 Sep;31(9):2135-41. doi: 10.1093/humrep/dew176. Epub 2016 Jul 4. PMID 27381766
- [Result] Sabra S, Malmqvist E, Saborit A, Gratacos E, Gomez Roig MD. Heavy metals exposure levels and their correlation with different clinical forms of fetal growth restriction. PLoS One. 2017 Oct 6;12(10):e0185645. doi: 10.1371/journal.pone.0185645. eCollection 2017. PMID 28985223
- [Result] Ovayolu A, Ovayolu G, Karaman E, Yuce T, Ozek MA, Turksoy VA. Amniotic fluid levels of selected trace elements and heavy metals in pregnancies complicated with neural tube defects. Congenit Anom (Kyoto). 2020 Sep;60(5):136-141. doi: 10.1111/cga.12363. Epub 2019 Nov 27. PMID 31743503

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-09): https://cdn.clinicaltrials.gov/large-docs/11/NCT04394611/Prot_SAP_000.pdf